CLINICAL TRIAL: NCT05041972
Title: A Global Phase 2 Study to Evaluate the Efficacy and Safety of ARX788 for Selected HER2-mutated or HER2-amplified/Overexpressed Solid Tumors
Brief Title: ARX788 in Selected HER2-mutated or HER2-amplified/Overexpressed Solid Tumors (ACE-Pan Tumor-02)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business strategy change
Sponsor: Ambrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-Pan tumor-02
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-04

CONDITIONS: HER2 Mutation-Related Tumors; HER2 Amplified Solid Tumors
Keywords: HER2 Mutation; HER2 Amplification; Non-Small Cell Lung Cancer (NSCLC); Colorectal (CRC); Biliary Tract Cancer (BTC); Breast Cancer; Other Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms; Breast Neoplasms | interventions — ARX788

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: HER2 Mutated Non-Small Cell Lung Cancer (NSCLC) (Experimental): Intervention: Drug: ARX788
  Interventions: Drug: ARX788
- Cohort 2: HER2 Mutation Breast Cancer (Experimental): Intervention: Drug: ARX788
  Interventions: Drug: ARX788
- Exploratory Cohort A: Other HER2-Mutated tumors (Experimental): Intervention: Drug: ARX788
  Interventions: Drug: ARX788
- Cohort 3: HER2 Amplification Biliary Tract Cancer (BTC) (Experimental): Intervention: Drug: ARX788
  Interventions: Drug: ARX788
- Cohort 4 HER2 Amplification Colorectal (CRC), Ovarian Endometrial, NSCLC, and other solid tumors (Experimental): Intervention: Drug: ARX788
  Interventions: Drug: ARX788
- Cohort 5: HER2 Mutation or HER2 Amplification Solid Tumors (Experimental): Intervention: Drug: ARX788
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — ARX788 will be administered by intravenous (IV) infusion every 3 weeks (Q3W).
  Other Names: ADC

SUMMARY:
A Global Phase 2 Study to Evaluate the Efficacy and Safety of ARX788 for Selected HER2-mutated or HER2-amplified/overexpressed Solid Tumors (ACE-Pan tumor-02)

DETAILED DESCRIPTION:
The study will enroll subjects with HER2-mutated or HER2-amplified/overexpressed locally advanced or metastatic solid tumor cancers whose prior standard of care therapies have failed. This basket trial will evaluate ARX788 across multiple cancer populations, as defined by HER2 genetic biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and older
* Life expectancy > 3 months
* Eastern Cooperative Oncology Performance Status ≤ 1
* HER2 status must be determined from a local Clinical Laboratory Improvement Amendments (CLIA) or equivalent-certified laboratory.
* Cohort 1, Cohort 2, and Explanatory Cohort A: HER2 mutated subjects with pre-specified HER2 activating mutation. Subjects with HER2 mutations in NSCLC (Cohort 1), breast cancer (Cohort 2), and other solid tumors (Cohort A) who have not received prior HER2 antibody drug conjugate (ADC) treatment are eligible.
* Cohort 3: Subjects with HER2 amplifications in biliary tract cancers (BTC) who have not received prior HER2 ADC treatment are eligible.
* Cohort 4: Subjects with HER2 amplifications in colorectal cancer (CRC), ovarian, endometrial, NSCLC and other solid tumors who have not received prior HER2 ADC treatment are eligible.
* Cohort 5 HER2 mutation or HER2 amplification: subjects with HER2 mutated or amplified tumors and have been previously treated with HER2 ADC are eligible.
* Subjects who are resistant or refractory to previous standard care of treatment.
* Subjects with stable brain metastases.
* Adequate organ functions.

Exclusion Criteria:

Any subject who meets any of the following criteria is excluded from the study:

* For Cohort 4: breast and gastric/GEJ cancer are excluded.
* Prior history of interstitial lung disease, pneumonitis, or other clinically significant lung disease within 12 months.
* History of ocular events, any current ongoing active ocular infections, or any chronic corneal disease unless approved by Medical Monitor.
* Exposure to any other investigational or commercial anticancer agents or therapies administered with the intention to treat malignancy within 14 days before the first dose of ARX788.
* Clinically significant surgical intervention (excluding diagnostic biopsy) within 21 days of the first dose of ARX788.
* Radiotherapy administered less than 21 days prior to the first dose of ARX788, or localized palliative radiotherapy administered less than 7 days prior to the first dose of ARX788, or radiotherapy-induced toxicity of Grade 2 or greater based on NCI-CTCAE v 5.0.

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of every 2 cycles (each cycle is 21 days)
  The confirmed objective response rate (ORR) of ARX788 by blinded independent central review (BICR) based on RECIST 1.1 in Cohorts 1-5.
  The ORR is defined as the number of subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of response evaluable subjects

SECONDARY OUTCOMES:
Duration of Response | 1 year
  DOR is defined as the time between the date of first response and the date of disease progression or death, whichever occurs first, will be computed for subjects with a BOR of CR or PR.
Best Overall Response (BOR) | At the end of every 2 cycles (each cycle is 21 days)
  BOR is defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Disease Control Rate (DCR) | 2 years
  DCR is defined as the proportion of complete response (CR), partial response (PR), and stable disease (SD) rates.
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time between date of first dose of study therapy and date of progression or death.
Overall Survival (OS) | 2 years
  Overall survival (OS) is defined as the time from first dose of study therapy to the date of death (any cause).
Time to Response (TTR) | At the end of every 2 cycles (each cycle is 21 days)
  Time to response (TTR) is defined as the time from the start of treatment to the first objective tumor response
Maximum serum concentration (Cmax) for ARX788, total antibody, and metabolites | Cycle 1 and Cycle 3
  Pharmacokinetic parameter maximum serum concentration (Cmax) for ARX788, total antibody, and metabolites.
Trough concentration (Ctrough) for ARX788, total antibody, and metabolites | Cycle 1 and Cycle 3
  Pharmacokinetic parameter trough concentration (Ctrough) for ARX788, total antibody, and metabolites.
Incidence of anti-drug antibodies (ADAs) | Predose at every cycle (each cycle is 21 days)
  Incidence of anti-drug antibodies (ADAs) following intravenous administration of ARX788 in participants with HER2-mutated or HER2-amplified locally advanced or metastatic solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Global Trial Lead, Study Director — Ambrx, Inc.
Locations (2):
- United States (2):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AMR Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available after the studies for which the medicine and indication have received marketing approval in European Union (EU) and United States (US) or regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.